CLINICAL TRIAL: NCT04859712
Title: A Diagnostic Test of Abnormal Sound Waves in Modern Pulsology of Lumbar Disc Herniation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, Professor, Qianfoshan Hospital
Other Study IDs: SFUYIN-03
Record Dates: First submitted 2021-03-14; First posted 2021-04-26 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2022-04

CONDITIONS: Lumbar Disc Herniation; Radial Artery
Keywords: Diagnostic Test; Lumbar Disc Herniation; Radial Artery
MeSH Terms: conditions — Intervertebral Disc Displacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trial group: 45 patients with lumbar disc herniation: The "Pulse Detection System of Sound Waves " was used to collect three parts and five layers of pulsed sound waves from the hands of 45 patients with lumbar disc herniation.
- Control group :45 relatively healthy people: The "Pulse Detection System of Sound Waves " was used to collect the three-parts and five-layers pulse sound waves of the hands of 45 relatively healthy people.

SUMMARY:
The purpose of this study is to use the " Pulse Detection System of Sound Waves " to collect the pulse information of recruited subjects, and to extract characteristic pulse information by multi-scale entropy, Fourier transform, Hilbert yellow transform, spectrum analysis, wavelet analysis and other methods. Evaluate the specificity, sensitivity, positive likelihood ratio and negative likelihood ratio of the "Pulse Detection System of Sound Waves" in the diagnosis of lumbar disc herniation.

DETAILED DESCRIPTION:
Pulse diagnosis is an important method to judge the status of patients in the process of diagnosis and treatment of traditional Chinese medicine. At present, the commonly used site of pulse diagnosis is the radial artery, which is divided into "cun", "guan" and "chi". Whether the diagnosis of lumbar disc herniation can be realized through pulse diagnosis has not been solved. Herniation of the lumbar intervertebral disc is a syndrome caused by degeneration of intervertebral disc, partial or complete rupture of the annulus fibrosus, protrusion of nucleus pulposus, or compression of nerve roots and cauda equina. In the area of compression, the blood supply is also limited to a certain extent, and the blood that should be in the normal laminar flow state gradually turns into a turbulent state, causing abnormal vibration, which is fused with a larger cluster of sound waves transmitted by the heart and then transmitted throughout the body. In this situation, the investigators can feel the combination of abnormal vibration waves by touching the pulse at different levels of the arteries near the surface of the body, including the radial artery. In long-term clinical practice, the investigators have found that the ulnar radial pulse of patients with lumbar disc herniation, i.e. the fifth layer of the ulnar radial pulse, often presents an unsmooth pulse. Therefore, the investigators believe that patients with lumbar disc herniation may have abnormal sound waves in the radial artery.

The investigators have found that there are low-frequency sound waves in the radial artery, which carry the physiological and pathological information of the organs in the body, and developed the "Pulse Detection System of Sound Waves". Previous projects have achieved certain results after exploring the abnormal sound waves of the radial artery in patients with sequelae of cerebral infarction, stable coronary heart disease, chronic gastritis and other diseases.

Therefore, this study will use the "Pulse Detection System of Sound Waves" to collect the sound waves in the radial artery of both hands from 45 patients with lumbar disc herniation and 45 relatively healthy people and carry out spectrum analysis and wavelet analysis to extract the pulse characteristics. The sensitivity and specificity of "Pulse Detection System of Sound Waves" in the diagnosis of lumbar disc herniation will be calculated. Supposed there are characteristic sound waves in the radial artery of patients with lumbar disc herniation, and these characteristic sound waves have some specific distributions, planes, and points that are different from the sound waves of relatively healthy persons. Then this study will explore and gradually confirm such characteristics and differences. It is expected to contribute to the pulse diagnosis of lumbar disc herniation.

ELIGIBILITY:
Inclusion Criteria:

- Trial group

1. Study time: March 9, 2021, to March 9, 2022 ;
2. Study site: The First Affiliated Hospital of Shandong First Medical University;
3. Patients with lumbar disc herniation who have not undergone lumbar surgery and who meet the diagnostic gold standard of symptoms, signs and imaging examinations should be comprehensively assessed.;
4. Patients who were first diagnosed with lumbar disc herniation less than 4 months ago;
5. Patients with a range of ages of 20-50 years and stable vital signs;
6. Patients who have informed consent to receive the pulse collection;

control group

1. Study time: March 9, 2021, to March 9, 2022 ;
2. Study site: The First Affiliated Hospital of Shandong First Medical University;
3. Relatively healthy people without lumbar disc herniation diagnosis;
4. Patients with a range of ages of 20-50 years and stable vital signs;
5. Patients who have informed consent to accept the pulse collection;

Exclusion Criteria:

- Trial group

1. Patients with lumbar spinal stenosis, lumbar tuberculosis, vertebral metastases, nerve root and cauda equina tumors, hip osteoarthropathy or aseptic necrosis of the femoral head, piriformis syndrome, ankylosing spondylitis, herpes zoster and other lumbar diseases;
2. Patients with diseases of the urinary system and reproductive system;
3. Patients who have undergone lumbar disc surgery;
4. Pregnant or lactating women;
5. Patients with other thoracic diseases;
6. Patients with gallbladder, pancreas and other diseases adjacent to the liver;
7. Patients with severe infectious diseases;
8. Those who are not easy to collect pulse manifestation such as pulse on back of wrist and oblique-running pulse;
9. Incomplete data due to subjective or objective reasons affect the judgment of results;
10. Patients with Parkinson's disease or other limb tremor;
11. Patients with atrial fibrillation.

control group

1. Patients with lumbar disc herniation;
2. Patients suffering from lumbar tuberculosis, ankylosing spondylitis and other serious diseases and difficult to maintain posture for a certain period of time;
3. Pregnant or lactating women;
4. Patients with severe infectious diseases;
5. Those who are not easy to collect pulse manifestation such as pulse on back of wrist and oblique-running pulse;
6. Incomplete data due to subjective or objective reasons affect the judgment of results;
7. Patients with Parkinson's disease or other limb tremor;
8. Patients with atrial fibrillation.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients with lumbar disc herniation and relatively healthy people
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2021-04-09 (Actual); Primary Completion 2022-04-25 (Estimated); Study Completion 2022-04-25 (Estimated)

PRIMARY OUTCOMES:
Frequencies of abnormal sound waves in the pulses. | The data will be collected, analyzed and calculated in about 7 days.
  Using the Pulse Detection System of Sound Waves (PDSSW) to collect the pulse waves of both hands. The percentage(%) of Frequencies of abnormal sound waves in the pulse will be calculated.
The changes of sound waves in the pulses. | The discovery of characteristic sound waves may take 3 months.
  The changes of sound waves at different Hertz (Hz) frequencies and SMPL amplitudes will be compared between patients with lumbar disc herniation and relatively healthy individuals.
Diagnostic test | Diagnostic tests may take about 1 month.
  The percentage (%) of specificity, sensitivity, positive likelihood ratio and negative likelihood ratio of the "Pulse Detection System of Sound Waves" in the diagnosis of patients with lumbar disc herniation.
Sound waves analysis | 1 month.
  The Hertz (Hz) of the different segments of the sound waves in Wavelet transform.
  The Hertz (Hz) of the different layers of the sound waves in Hilbert-Huang. The SMPL amplitudes of the sound waves in Discrete Fourier Transform. The sampEn of sound waves in Sample Entropy.

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Song, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Background] Rickers KW, Pedersen PH, Tvedebrink T, Eiskjaer SP. Comparison of interventions for lumbar disc herniation: a systematic review with network meta-analysis. Spine J. 2021 Oct;21(10):1750-1762. doi: 10.1016/j.spinee.2021.02.022. Epub 2021 Mar 3. PMID 33667683
- [Background] Ishitani H, Tamura T, Kanaya S, Fujimoto H. Examination of the regression model to quantify the degree of low back pain and lower limb symptoms in patients with lumbar disc herniation by the Japanese Orthopaedic Association Back Pain Evaluation Questionnaire (JOABPEQ). PLoS One. 2020 Dec 14;15(12):e0243861. doi: 10.1371/journal.pone.0243861. eCollection 2020. PMID 33315945
- [Background] Siccoli A, Schroder ML, Staartjes VE. Association of age with incidence and timing of recurrence after microdiscectomy for lumbar disc herniation. Eur Spine J. 2021 Apr;30(4):893-898. doi: 10.1007/s00586-020-06692-1. Epub 2020 Dec 14. PMID 33315158
- [Background] Bilton K, Hammer L, Zaslawski C. Contemporary Chinese pulse diagnosis: a modern interpretation of an ancient and traditional method. J Acupunct Meridian Stud. 2013 Oct;6(5):227-33. doi: 10.1016/j.jams.2013.04.002. Epub 2013 Apr 24. PMID 24139459
- [Background] Shimony N, Louie C, Barrow D, Osburn B, Noureldine MHA, Tuite GF, Carey CM, Jallo GI, Rodriguez L. Adolescent Disc Disease: Risk Factors and Treatment Success-Related Factors. World Neurosurg. 2021 Apr;148:e314-e320. doi: 10.1016/j.wneu.2020.12.126. Epub 2021 Jan 4. PMID 33412329

DOCUMENTS (1):
  • Informed Consent Form (2021-02-28): https://cdn.clinicaltrials.gov/large-docs/12/NCT04859712/ICF_000.pdf